CLINICAL TRIAL: NCT07049432
Title: A Phase I Study of N-803 Maintenance Therapy Following CD19 Directed CAR T-cell Therapy in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphomas (CARMEN-803 Trial)
Brief Title: N-803 Maintenance Therapy Post CAR T-cell Therapy in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphomas
Acronym: CARMEN-803
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCI189957
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-06

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-803 (Experimental): Participants receive N-803 subcutaneously (SubQ) administered on day 1 of each 21-day cycle for up to 6 cycles.
  Interventions: Drug: N803

INTERVENTIONS:
Drug: N803 — N-803 subcutaneously (SubQ) administered on day 1 of each 21-day cycle for up to 6 cycles.

SUMMARY:
The purpose of this clinical trial is to learn whether the study drug N-803 is safe and tolerable in patients with B-cell non-Hodgkin lymphoma who have undergone CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Subjects with histologically confirmed B-cell NHL who have received commercially approved CD19-directed CAR T-cell therapy per FDA label
* Subjects achieving CR or PR per Lugano Criteria to CAR T-cell therapy on D+30 post-CAR-T.
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥750 cells/mm3 (≥0.75 x 10^9/L) independent of G-CSF support
    * Platelet count ≥50,000 cells/mm^3 (≥50 x 10^9/L) independent of transfusion support
    * Hemoglobin ≥ 7 g/dL (≥ 70 g/L) independent of transfusion support
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) or ≤ 3x ULN with Gilbert's disease.
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Subjects with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:

      * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
      * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy, or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 6.4.1.
* CRS and ICANS grade 0 at the time of enrollment and N-803 injection. Subjects must be off steroids and ≥7 days from tocilizumab or other anti-cytokine agent administration.
* Clinically significant adverse effects from any prior treatment (e.g. prior surgery, radiotherapy, or other antineoplastic therapy) must have resolved or have been determined to be clinically stable per the Investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior therapy with N-803, IL-2 or IL-15 based therapy.
* Receiving other investigational agents.
* Any ongoing toxicity from CAR T-cell therapy that, in the judgment of the investigator, may interfere with study treatment.
* Autoimmune disease requiring active treatment, other than corrected hypothyroidism and diabetes mellitus type 1.
* History of a prior or current malignancy that, in the opinion of the investigator, is likely to negatively impact subject participation or safety.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  -- Cardiovascular disorders:
  * Stroke or intracranial hemorrhage within 6 months of enrollment
  * Unstable angina or acute coronary syndrome within the past 2 months prior to study enrollment
  * History of myocardial infarction within 3 months prior to study enrollment in the 12 months prior to study enrollment
  * ≥ Grade 3 NYHA functional classification system of heart failure, uncontrolled or symptomatic arrhythmias
  * Left ventricular ejection fraction < 40% in the 12 months prior to study enrollment.

    ---- Note: A screening echo is not required for enrollment.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known HIV infection.
* Active infection including hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  -- Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal, or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and medical monitor may pose a risk for patient participation. Screening for chronic conditions is not required.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 7.7. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of N-803 post CAR T-cell therapy | 4 years
  determination of a dose level for the phase 2 study (RP2D)
Determination of a dose level for the phase 2 study (RP2D) of N-803 post CAR T-cell Therapy | 4 years
  determination of a dose level for the phase 2 study (RP2D)

SECONDARY OUTCOMES:
The proportion of patients with a Partial Response (PR), per Lugano criteria, who achieve a Complete Response (CR) by the end of Cycle 6. | 2 years
  To assess the rate of conversion from PR to CR at the end of Cycle 6.
Duration of response (DoR), defined as the interval of time from the date of initial documented response (PR or CR per Lugano criteria) to the time of progression, the start of a new therapy, or death from any cause. | 2 years
  To assess the DOR
Progression-free survival (PFS) as defined as the time from study drug initiation to the time documented disease progression (as assessed by Lugano Criteria) or death from any cause. | 2 years
  To assess median and 2-year PFS
Overall survival (OS) as defined as the time from initiation of study therapy until death from any cause. | 2 years
  To assess median and 2-year OS

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States